CLINICAL TRIAL: NCT03962400
Title: Randomized Trial of Reinforcement Learning for the Dosing of Warfarin
Brief Title: Reinforcement Learning for Warfarin Dosing
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study did not receive anticipated funding and therefore never opened to enrollment. The study was never submitted to the IRB for approval since the funding failed.
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Adam Edward Gaweda, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KDP002
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Clotting Disorder
Keywords: warfarin
MeSH Terms: conditions — Hemostatic Disorders | interventions — Reinforcement Machine Learning

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial of 2 groups. Subjects in the Control group will receive warfarin with dose adjustment guided by standard protocol. Subjects in the Treatment group will receive warfarin with dose adjustment guided by personalized protocol.
Who Masked: Participant
Masking Description: Subjects will not be informed of group designation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Subjects will have warfarin dose determined in the usual fashion by a health care provider.
  Interventions: Procedure: Heath Care Provider
- Treatment (Experimental): Subjects will have warfarin dose determined using a reinforcement learning computer model.
  Interventions: Procedure: Reinforcement Learning

INTERVENTIONS:
Procedure: Reinforcement Learning — New computer based procedure for determining dose using a decision support tool
  Arms: Treatment
Procedure: Heath Care Provider — Warfarin dose will be determined by a qualified health care provider
  Arms: Control

SUMMARY:
This is a clinical study designed to test the hypothesis that a computer model for dosing warfarin is superior to current clinical practice. Subjects will be randomized to two groups based on how warfarin dose is determined and followed for 6 months. The primary outcome is the percent of the time that the INR is maintained in the effective range.

DETAILED DESCRIPTION:
This will be a single-center, open-label, randomized prospective study. Primary outcome will be percent of time within a specific INR range. Subjects will be randomized to to control and treatment groups and stratified 1:1 based on sex. The control group will have warfarin doses adjusted by experts in the treatment of patients with warfarin. The treatment group will have warfarin doses determined using a clinical support tool based on reinforcement learning. Based on simulations of the experimental design with an expectation that the percent of INR values within the target range increase by 20%, 70 subjects per group are required for statistical significance. Based on an attrition rate of 15%, the investigators will enroll 80 subjects per group. Statistical analysis will compare the percent of patients within the target INR range between groups as the primary outcome with number of adverse events between groups as the safetly outcome.

ELIGIBILITY:
Inclusion Criteria:

* Receiving anticoagulation treatment with warfarin.

Exclusion Criteria:

* Pregnancy.

  * History of hemorrhagic cerebrovascular incident.
  * Acquired or inherited hemophilia.
  * Thrombocytopenia (<100,000 platelets per mm3) on 2 occasions separated by 2 days.
  * Anemia with hemoglobin concentration < 10 g/dL.
  * Active cancer excluding non-melanoma skin cancers.
  * Active liver disease as documented by prolonged baseline INR ≥ 1.6.
  * Uncontrolled hypertension with 2 readings >180/110.
  * Recent (< 2 weeks) neurosurgical procedure.
  * Enrollment in hospice program for any diagnosis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent in Range | 6 months
  Percent of INR measurements within the Target Range

SECONDARY OUTCOMES:
Adverse Events | 6 Months
  Composite of all adverse events attributed to warfarin

IPD SHARING:
Plan to Share IPD: No